CLINICAL TRIAL: NCT05178446
Title: The New Onset of GERD After Sleeve Gastrectomy: a Systematic Review
Brief Title: GERD After Sleeve Gastrectomy
Status: Completed | Type: Observational
Sponsor: University of Foggia (Other)
Responsible Party: Principal Investigator, Giovanna Pavone, Medical Doctor, University of Foggia
Other Study IDs: 3
Record Dates: First submitted 2021-12-12; First posted 2022-01-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Morbid Obesity; GERD
MeSH Terms: conditions — Obesity, Morbid; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main adverse effect is gastroesophageal reflux disease (GERD), with concern on the development of Barrett's esophagus and esophageal adenocarcinoma in the long term. However, the relationship between SG and GERD is complex. The aim of this study is to systematically evaluate all published data existing in the literature to evaluate the effect of sleeve gastrectomy on GERD, esophagitis, BE in order to clarify the long-term clinical sequelae of this procedure.

This systematic review was conducted in accordance with the guidelines for Preferred Reporting Items for Systematic Review and Meta-analyzes (PRISMA).

Published studies that contained outcome data for primary sleeve gastrectomy associated with the primary and secondary outcomes listed below were included.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent to sleeve gastrectomy with reflux symptoms

Exclusion Criteria:

* Patients underwent to other bariatric procedures

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Obese patients underwent to sleeve gastrectomy with GERD symptoms
Sampling Method: Probability Sample
Enrollment: 14362 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Gastroesophageal reflux disease after bariatric surgery | from 2014 to 2018
  Number of patients underwent sleeve gastrectomy with GERD

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Tartaglia, Study Director — University of Foggia
Locations (1):
- University of Foggia, Foggia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pavone G, Tartaglia N, Porfido A, Panzera P, Pacilli M, Ambrosi A. The new onset of GERD after sleeve gastrectomy: A systematic review. Ann Med Surg (Lond). 2022 Apr 5;77:103584. doi: 10.1016/j.amsu.2022.103584. eCollection 2022 May. PMID 35432994

DOCUMENTS (1):
  • Study Protocol (2021-12-14): https://cdn.clinicaltrials.gov/large-docs/46/NCT05178446/Prot_000.pdf